CLINICAL TRIAL: NCT03494062
Title: Exercise in Juvenile Takayasu Disease: a Randomized Controlled Trial
Brief Title: Exercise in Juvenile Takayasu Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Takayasu&Exercise
Record Dates: First submitted 2018-03-05; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Takayasu's Arteritis
MeSH Terms: conditions — Takayasu Arteritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Home-based exercise intervention
  Interventions: Behavioral: Exercise
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Exercise — Home-based exercise training
  Arms: Exercise

SUMMARY:
Juvenile Takayasu disease is characterized by chronic inflammation that leads to vascular disease. Exercise may render anti-inflammatory effects and protect against cardiovascular events. This trial aims to investigate the therapeutic role of exercise in juvenile Takayasu disease.

DETAILED DESCRIPTION:
Takayasu's Arteritis (TA) is a chronic inflammatory disease that affects large and medium-sized arteries. The number of cases describe in children and adolescents has growing, and the hypertension is one of the symptoms most common, followed by other manifestations that affects cardiovascular systems. All clinical manifestations may aggravate by physical inactivity and can creating a vicious cycle of inflammation, whereas the risks of morbidity and mortality increase significantly in the pediatric population, impairing function and physical capacity, quality of life and evolution to adult life. Thereby, physical exercise it is show to be an efficient strategy to reduce all these risk factors, however, no one study, until now, was conducted to available the effects of exercise in children with TA. Objective: Investigated the effects of 12-week home-based exercise program, where the patients receive a guideline from a physical education professional, teaching how to do the exercise at home. The beneficial effects of the programs expect is to be associated with improved cardiovascular risk factors, function and physical capacity, and body composition. Methods: This is a prospective, longitudinal and randomized clinical trial. All patients will be recruited at the Clinical Hospital of the University of Sao Paulo Medical School (HC-FMUSP), in the Laboratory of Evaluation and Conditioning in Rheumatology, Pediatric Rheumatology outpatient clinics of the Department of Pediatrics, Federal University of São Paulo and The Children's Institute of the University of São Paulo and the Vasculitis Unit of the HC-FMUSP Rheumatology Service. In order to evaluate the therapeutic effects of exercise program act on TA, the following pre and post intervention evaluations will be performed: physical activity level; Global clinical evaluation; Anthropometry and body composition; Hematological and inflammatory blood parameters; Cardiovascular risk factors; Aerobic capacity; Functional capacity and fatigue; quality of life; and 18 FDG PET with magnetic resonance angiography.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of juvenile Takayasu disease

Exclusion Criteria:

* cardiac and renal insufficiency
* physical limitation hampering exercise training
* non-controlled metabolic disorders
* associated chronic diseases (last 6 months)

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Arterial inflammation | 12 weeks
  as assessed by positron emission tomography - magnetic ressonance (PET-MR)
Blood inflammatory markers | 12 weeks
  interleukin-6, interleukin 10, interleukin-12
Blood inflammatory marker | 12 weeks
  C-reactive protein
velocity sedimentation rate | 12 weeks
  velocity sedimentation rate

SECONDARY OUTCOMES:
Maximal aerobic capacity | 12 weeks
  as assessed by maximal cardiopulmonary test
Body composition | 12 weeks
  Lean, fat and bone mass, as assessed by dual energy x-ray absorptiometry
Timed stands test | 12 weeks
  The test is performed by measuring the time to stand up and down for 30 seconds. The patient should make two attempts and the best performance will be considered for the analyzes.
timed-up-and-go test | 12 weeks
  The "Timed Up-And-Go" test, which evaluates the time it takes for the patient to get up from a chair, walk three meters, make a 180-degree turn, and return to the chair. The patient should perform two attempts and the best performance will be considered for the analyzes.
Isometric strength | 12 weeks
  handgrip test
Maximal strength test | 12 weeks
  will be performed by the maximum repetition test, where the objective is to find a maximal repetition for lower limbs by leg press exercise 45º and for upper limbs by bench press exercise
The Paediatric Vasculitis Activity Score (PVAS) | 12 weeks
  The final PVAS is a clinical index of 64 manifestations of active vasculitis, divided into five domains: general, cutaneous, cardiovascular, abdominal and renal.
National Institute of Health (NIH) | 12 weeks
  The NIH criteria is an instrument that will evalueted the disease specific symptoms and his activity. Active disease will arbitrarily defined as new onset or worsening of at least 2 of the following 4 features: (I) signs and symptoms of vascular ischemia or inflammation (e.g. claudication, decreased or absent extremity pulses or blood pressure, bruits, or carotidynia); (2) elevated erythrocyte sedimentation rate; (3) angiographic abnormalities; and (4) systemic symptoms not attributable to another disease.
Indian Takayasu's Arteritis Activity Score 2010 (ITAS2010 | 12 weeks
  ITAS2010 contains 44 items with 33 features arising from the cardiovascular system. Seven key items are weighted to score 2 and all others score 1 only.
Childhood Health Assessment Questionaire (CHAQ) | 12 weeks
  The Childhood Health Assessment Questionnaire (CHAQ) is a disease specific health instrument that measures functional ability in daily living activities in children
Physical activity levels | 12 weeks
  The level of physical activity of patients will be measured using the Actigraph GT3x® triaxial accelerometer (Actigraph®).
Fatigue severity scale FSS | 12 weeks
  The Fatigue severity scale will be used to monitor the change in fatigue in response to the intervention. For each item, you must tick from 1 totally disagree to 7 agree totally. The total number of points may vary from 9 to 63, and it is established that values equal to or greater than 28 are indicative of the presence of fatigue
Quality of life | 12 weeks
  as assessed by Short-Form-36
Hypotension after acute exercise session | 12 weeks
  after maximal aerobic capacity, the blood pressure will be will be measured in the four limbs, both arms and legs, every fifteen minutes, for an hour.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BG Gualano, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Castanho, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Astley C, Clemente G, Terreri MT, Carneiro CG, Lima MS, Buchpiguel CA, Leao Filho H, de Sa Pinto AL, Silva CA, Campos LMA, Aikawa NE, Gil S, Pereira RMR, Roschel H, Gualano B. Home-Based Exercise Training in Childhood-Onset Takayasu Arteritis: A Multicenter, Randomized, Controlled Trial. Front Immunol. 2021 Jul 28;12:705250. doi: 10.3389/fimmu.2021.705250. eCollection 2021. PMID 34394103